CLINICAL TRIAL: NCT03721770
Title: Psychological Impact in a Relative, Following the Announcement of the Death of a Loved One After Cardiac Arrest and the Early Request for Organ Donation: an Observational, Prospective Study
Brief Title: Psychological Impact in a Relative, Following the Announcement of the Death of a Loved One After Cardiac Arrest and the Early Request for Organ Donation
Acronym: REPERPSY
Status: Completed | Type: Observational
Sponsor: frederic ADNET (Other)
Responsible Party: Sponsor-Investigator, frederic ADNET, MD, PhD, Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence
Organization: Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence (Other)
Other Study IDs: LIC16160108
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Post Traumatic Stress Disorder; Family; Psychological Distress; Organ and Tissue Procurement
Keywords: organ donation; family; Post Traumatic Stress Disorder; Bereavement
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relatives: Relative or adult companion (age <18 years) of a patient who died of cardiac arrest after organ removal request. A parent is defined as a close relative of the first degree: husband-wife, father-mother, son-daughter. Only one loved one is included per patient. Inclusion order of priority is husband-wife / father-mother / son-daughter.

SUMMARY:
The fight against the scarcity of grafts is a major public health issue in France. Despite a very good success rate of transplants from brain-dead donors or living donors, the waiting time for transplantation continues to increase, leading to morbidity and mortality, as well as medical costs. Since 2005, the BioMedicine Agency has implemented a protocol authorizing kidney and liver samples taken from deceased donors after cardiac arrest (DDAC). This type of sampling has become a common practice in several regions of France and Europe. In case of DDAC, the sampling protocol poses a significant temporal constraint, since the patient must be taken within 6 hours after the cardiac arrest. This constraint leads to a specific organization of the announcement of the death and the request for non-opposition to the levy.

The brutal loss of a loved one is a potentially traumatic experience for family members. The manifestations of the pathological components of mourning such as post-traumatic stress disorder, anxio-depressive syndrome, pathological bereavement, are often expressed early in the first year after the death of the loved one. Families of organ donor patients probably represent a population at high risk for the expression of psychiatric conditions such as post-traumatic stress disorder or pathological bereavement. The limited time available to prepare relatives to make a decision could promote the expression of psychiatric morbidity in the short or medium term. The data on this new transplantation procedure and its psychological consequences are insufficient, and we consider that if a state of post-traumatic stress occurred in more than 50% of parents, the procedure of announcement would be reviewed. The purpose of this study is to test this hypothesis.

Most of the work on relatives of potential organ donors has focused on procedures for brain death. Most of this work has focused on characterizing the determinants of acceptance or refusal of organ donation in the family. The literature relating to the follow-up of relatives of a patient after organ donation is very poor: very few studies have focused on the psychological consequences and / or the psychological state of this population in the period post-death. In addition, very few qualitative and quantitative studies make it possible to evaluate the appearance of psychopathological manifestations related to the announcement of death simultaneously with a request for organ removal. This research, therefore, will make it possible to estimate the possible psychological impact on the bereaved family as well as an assessment of the psychological state. A mixed methodology (quantitative and qualitative) will make it possible to highlight explanatory factors of the quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* Parent or adult companion of a patient who died of cardiac arrest after organ removal (Inclusion order of priority is husband-wife / father-mother / son-daughter)
* Only one loved one is included per patient.

Exclusion Criteria:

* Age < 18 years
* Refusal to participate in the study
* Difficulty in communication (foreign, language, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The relatives will be recruited during the interview with the coordination team of organs and tissues, after acceptance or refusal of organ donation.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Score ≥ 33 on the Impact of Event Scale - Revised. | 3 months
  Percentage of relatives with post-traumatic stress disorder at 3 months with a score ≥ 33 on the Impact of Event Scale - Revised.
  The Impact of Event Scale - Revised measures symptoms of intrusion, avoidance, numbing and hyperarousal with respect to a particular life-threatening event. Subscales of the scale: Intrusion scale (range 0-24 score); avoidance scale (range 0-26 score); hyperarousal scale (range 0-18 score. Range of the scale 0-88 scores.
  Score 24 and more: PTSD is a clinical concern. Score 33 and above : This represents the best cutoff for a probable diagnosis of PTSD Score 37 and more : This is high enough to suppress the immune system's functioning (even 10 years after an impact event).

SECONDARY OUTCOMES:
Post Traumatic Stress Disorder Diagnosis And Major Depressive Episode Diagnosis (Mini International Neuropsychiatric Interview - Version 5.0.0 Module I. Post Traumatic Stress Disorder and Module A. Major Depressive Episode) | 3 months et 1 year
  Psychological Assessment of Post Traumatic Stress Disorder Diagnosis and Major Depressive Episode Diagnosis.
Score of depression and anxiety (Hospital of Anxiety and Depression Scale). | 3 months and 1 year
  Hospital of Anxiety and Depression Scale measures an anxio-depressive symptomatology and evaluates its severity. It does not try to distinguish different types of depression or anxiety states. This scale was constructed excluding any item concerning somatic aspects. Subscale anxiety (range score 0-21) and Subscale depression (range score 0-21). The thresholds for the sub scores are:
  0-7 score = no anxiety disorder or depressive disorder; 8-10 = anxiety disorder or depressive disorder suspected; 11-21 = anxiety disorder or depressive disorder.
  Range total score= 0-42. The thresholds for a total score are:
  0-14 score= no anxiety or depressive disorder 15-42 score= existence of an anxiety or depressive disorder.
Score of pathological mourning (Inventory of Complicated Grief) | 1 year
  Inventory of Complicated Grief measures the symptoms of 'complicated grief'.The complicated grief is identified by the extended length of time of the symptoms, the interference in normal function caused by the symptoms, or by the intensity of the symptoms (for example, intense suicidal thoughts or acts).The complicated grief may appear as a complete absence of grief and mourning, an ongoing inability to experience normal grief reactions, delayed grief, conflicted grief, or chronic grief. Factors that contribute to the chance that one may experience complicated grief include the suddenness of the death, the gender of the person in mourning, and the relationship to the deceased.
  Range total score= 0-88. Respondents with ICG scores greater than 25 are significantly more impaired in social, general, mental and physical health functioning and in bodily pain than those with ICG scores less than or equal to 25.
  No subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- ADNET Frederic, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Background] Dominguez-Gil B, Haase-Kromwijk B, Van Leiden H, Neuberger J, Coene L, Morel P, Corinne A, Muehlbacher F, Brezovsky P, Costa AN, Rozental R, Matesanz R; European Committee (Partial Agreement) on Organ Transplantation. Council of Europe (CD-P-TO). Current situation of donation after circulatory death in European countries. Transpl Int. 2011 Jul;24(7):676-86. doi: 10.1111/j.1432-2277.2011.01257.x. Epub 2011 Apr 19. PMID 21504489
- [Background] Fieux F, Losser MR, Bourgeois E, Bonnet F, Marie O, Gaudez F, Abboud I, Donay JL, Roussin F, Mourey F, Adnet F, Jacob L. Kidney retrieval after sudden out of hospital refractory cardiac arrest: a cohort of uncontrolled non heart beating donors. Crit Care. 2009;13(4):R141. doi: 10.1186/cc8022. Epub 2009 Aug 28. PMID 19715564
- [Background] Eckenrod EL. Psychological/emotional trauma of donor families. Transplant Proc. 2008 May;40(4):1061-3. doi: 10.1016/j.transproceed.2008.03.048. PMID 18555115